CLINICAL TRIAL: NCT06784882
Title: A Pilot Randomized Controlled Trial Assessing Pain and Opioid Outcomes Among Patients Undergoing Total Knee Arthroplasty Receiving 5-Day Outpatient Adductor Canal Continuous Versus Single Injection Blocks
Brief Title: Continuous Versus Single Injection Adductor Canal Blocks for Outpatient Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rodney Gabriel, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 811228
Record Dates: First submitted 2025-01-11; First posted 2025-01-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Postoperative Pain; Surgery
Keywords: regional anesthesia; total knee arthroplasty; nerve block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous adductor canal block (Experimental): single injection with ropivacaine (0.5%) of the adductor canal block and a 5-day continuous perineural infusion of ropivacaine (0.2%) (experimental group)
  Interventions: Device: continuous peripheral nerve block with OnQ pump
- single injection adductor canal block (Active Comparator): single injection with ropivacaine (0.5%) of the adductor canal block and no continuous nerve block added
  Interventions: Drug: single injection nerve block

INTERVENTIONS:
Device: continuous peripheral nerve block with OnQ pump — For continuous nerve blocks, the infusion pump that will be used are OnQ pumps (Avanos, Alpharetta, GA) and pre-filled with ropivacaine 0.2% and provided by UCSD's Investigational Drug Services.
  Arms: Continuous adductor canal block
Drug: single injection nerve block — An adductor canal single injection nerve block will be performed per standard of care. The adductor canal will be identified by ultrasound in the short-axis view. The distal aspect of the femoral triangle (and beginning of the adductor canal) will be identified distal to the mid-thigh in the ipsilateral limb. Using ultrasound guidance, a standard Tuohy block needle will be advanced through a skin wheal of lidocaine until its tip is in the hypoechoic area immediately distal saphenous nerve adjacent to the femoral artery. Twenty milliliters of ropivacaine 0.5% will be injected in divided doses with repeated negative aspiration.
  Arms: single injection adductor canal block

SUMMARY:
This is a single-center pilot study to determine if an adductor canal continuous nerve block is superior to single injection nerve block following total knee arthroplasty. Investigators will randomize participants to either continuous nerve block or single injection nerve block for the adductor canal preoperatively. They will assess differences in pain (measured in numeric rating scale), opioid consumption, and physical therapy milestones from postoperative day 0 to 7.

DETAILED DESCRIPTION:
Adductor canal blocks are standard care for postoperative analgesia following total knee arthroplasty. Adductor canal blocks involve depositing local anesthetic (ropivacaine) around the saphenous nerve at the location of the adductor canal on the ipsilateral thigh. At UCSD, the standard care is to perform single injection adductor canal blocks for research participants undergoing total knee arthroplasty prior to surgery in the preoperative waiting area.

Participants will be randomized to either: (1) single injection with ropivacaine (0.5%) of the adductor canal block AND a 5-day continuous perineural infusion of ropivacaine (0.2%) (experimental group); versus (2) single injection with ropivacaine (0.5%) of the adductor canal block and no continuous nerve block added.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants of at least 18 years of age
2. Undergoing a primary, unilateral, total knee arthroplasty
3. Planned single-injection adductor canal nerve block
4. Weight > 50 kg (to minimize the risk of local anesthetic toxicity)

Exclusion Criteria:

1. chronic opioid or tramadol use: daily oxycodone equivalents > 20 mg for > 4 weeks
2. neuro-muscular deficit of the surgical limb
3. moderate pain (NRS > 3) in an anatomic location other than the surgical site
4. planned hospital admission following surgery
5. history of opioid misuse
6. those who lack capacity to complete informed consent
7. inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access)
8. incarceration
9. pregnancy
10. allergy to amide local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
analgesic effect of 5-day continuous nerve block of the adductor canal relative to a single inection nerve block with ropivacaine. | 7 days
  Numeric Rating Scale (NRS) for pain will be superior daily with continuous adductor canal blocks on postoperative days 1-7 following total ankle arthroplasty as compared with single-injection adductor canal blocks (as measured by the "average" daily NRS within the Brief Pain Inventory)
opioid consumption of 5-day continuous nerve block of the adductor canal relative to a single inection nerve block with ropivacaine. | 7 days
  Opioid consumption will be superior daily with continuous adductor canal blocks on postoperative days 1-7 following total ankle arthroplasty as compared with single-injection adductor canal blocks (measured in oxycodone equivalents)

SECONDARY OUTCOMES:
physical and emotional functioning of 5-day continuous nerve blocks relative to a single injection nerve blocks with ropivacaine | 7 days
  The physical and emotional functioning of research participants will be superior daily with continuous adductor canal blocks on postoperative days 1-7 following total ankle arthroplasty as compared with single-injection adductor canal blocks (as measured with the Brief Pain Inventory Interference Subscale)
improvement in physical therapy milestones of 5-day continuous nerve blocks relative to a single injection nerve blocks with ropivacaine | 30 days
  Knee injury and osteoarthritis outcome score for joint replacement (KOOS JR)
30-day pain score measured in Numeric Rating Scale | 30 days
  At around 30 days postoperatively, the patients average pain score measured in the numeric rating scale (0-10) will be assessed.
30-day postoperative opioid consumption | 30 days
  Around 30 days postoperatively, the average opioid consumption will be assessed. This will be based on the average opioid consumption over the preceding week at 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847